CLINICAL TRIAL: NCT03255356
Title: International Multicentre Observational Trial of Perioperative Ventilatory Management in Cardiac Surgery
Brief Title: Ventilation in Cardiac Surgery
Acronym: VENICE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 16-081
Record Dates: First submitted 2017-06-12; First posted 2017-08-21 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-03

CONDITIONS: Respiratory Complication; Respiration, Artificial; Anesthesia, General; Bypass, Cardiopulmonary
Keywords: Postoperative pulmonary complications; Protective mechanical ventilation; Alveolar lung recruitment manoeuvres; Cardiac Surgery Procedures
MeSH Terms: conditions — Respiratory Aspiration | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: An anonymised questionnaire will be answered for each includable consecutive patient after verifying the absence of exclusion criteria.
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — An anonymised questionnaire will be answered for each includable consecutive patient after verifying the absence of exclusion criteria.
  Other Names: not adapted

SUMMARY:
The purpose of this study is to evaluate prospectively ventilatory practices in the perioperative cardiac surgery period.

DETAILED DESCRIPTION:
This is a International Multicentre Observational Trial on all adult cardiac surgery patients with cardiopulmonary bypass (CPB).

ELIGIBILITY:
Inclusion Criteria:

* All consecutive cardiac surgery patients with CPB during one predefined period,
* Elective or urgent surgery as defined by EuroSCORE2.

Exclusion Criteria:

* Refusal of consent,
* Pregnant women,
* Age < 18 years,
* Heart transplant, ECLS, ventricular assist
* Emergency or salvage surgery as defined by EuroSCORE2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult cardiac surgery patients with cardiopulmonary bypass (CPB).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
incidence of use prophylactic protective mechanical ventilation defined with with low tidal volume (6 to 8 ml / kg based on the ideal body weight) | 1 day
  percent

SECONDARY OUTCOMES:
incidence of using positive end-expiratory pressure | 1 day
  (PEEP)> 5 cmH2O
incidence of using at least 2 alveolar lung recruitment manoeuvres | 1 day
  percent
incidence of using a protective ventilation bundle combining prophylactic protective mechanical ventilation and at least 2 alveolar recruitment manoeuvres | 1 day
  percent
incidence of postoperative pulmonary complications | 1 month postoperatively
  percent

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Olivier Fischer, MD, PhD, Principal Investigator — University Hospital of Caen
Locations (10):
- CUB Erasm, Université libre de Bruxelles, Brussels, Belgium
- Universidade Federal de São Paulo (UNIFESP), Brasil, Brazil
- General University Hospital, Prague, Czechia
- Caen University Hospital, Caen, France
- Klinik für Anästhesiologie und Intensivmedizin, Jena, Germany
- Azienda Ospedaliera Universitaria, Pisa, Italy
- Osaka city University Graduate school of Medecine, Ōsaki, Japan
- VU University Hospital, Amsterdam, Netherlands
- St Olav University Hospital, Trondheim, Norway
- Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] Lellouche F, Delorme M, Bussieres J, Ouattara A. Perioperative ventilatory strategies in cardiac surgery. Best Pract Res Clin Anaesthesiol. 2015 Sep;29(3):381-95. doi: 10.1016/j.bpa.2015.08.006. Epub 2015 Sep 4. PMID 26643102
- [Background] Guldner A, Kiss T, Serpa Neto A, Hemmes SN, Canet J, Spieth PM, Rocco PR, Schultz MJ, Pelosi P, Gama de Abreu M. Intraoperative protective mechanical ventilation for prevention of postoperative pulmonary complications: a comprehensive review of the role of tidal volume, positive end-expiratory pressure, and lung recruitment maneuvers. Anesthesiology. 2015 Sep;123(3):692-713. doi: 10.1097/ALN.0000000000000754. PMID 26120769